CLINICAL TRIAL: NCT01727921
Title: Endoscopic Ultrasound-guided Fine Needle Tissue Acquisition With 22- and 25-gauge ProCore Needle in Solid Pancreatic and Peripancreatic Masses: A Prospective Comparative Study
Brief Title: Comparative Study of 22 and 25 Gauge ProCore EUS-guided Biopsy in Pancreatic Mass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Kwang Hyuck Lee, Assistant Professor of Medicine, Division of Gastroenterology, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2012-08-066-001
Record Dates: First submitted 2012-10-21; First posted 2012-11-16 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Pancreatic Neoplasms
Keywords: ProCore FNA biopsy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 22 gauge ProCore needle biopsy (Active Comparator): EUS-guided pancreatic or peripancreatic mass biopsy with 22 gauge ProCore biopsy needle.
  Interventions: Device: 22 gauge ProCore needle biopsy
- 25 gauge ProCore needle biopsy (Active Comparator): EUS-guided pancreatic or peripancreatic mass biopsy with 25 gauge ProCore biopsy needle.
  Interventions: Device: 25 gauge ProCore needle biopsy

INTERVENTIONS:
Device: 22 gauge ProCore needle biopsy — 22 gauge, EchoTip® ProCore™ High Definition Ultrasound Biopsy Needle
  Arms: 22 gauge ProCore needle biopsy
Device: 25 gauge ProCore needle biopsy — 25 gauge, EchoTip® ProCore™ High Definition Ultrasound Biopsy Needle
  Arms: 25 gauge ProCore needle biopsy

SUMMARY:
Background:

EUS-guided fine needle aspiration (FNA) is a major diagnostic tool in the patient with pancreatic mass with high specificity, specificity and accuracy. However FNA with small needle has sometimes failed in acquisition of tissue due to small caliber. To overcome this limitation, newly designed ProCore needle was developed and flexible 22 and 25 gauge ProCore needles were frequently used. However there was no comparative study of the efficacy and accuracy between 22 and 25 gauge ProCore needle yet.

Aim:

To compare the efficacy and accuracy of EUS-guided FNA between 22 and 25 gauge ProCore needle. (The investigators hypothesized that the accuracy of 25 gauge Procore needle is not inferior to 22 gauge ProCore needle.)

DETAILED DESCRIPTION:
Patient and methods:

Patients who have pancreatic or peripancreatic mass in imaging studies which need pathologic confirm. These patients were randomly assigned to 22 gauge or 25 gauge group.

Procedure:

They underwent EUS-guided FNA, 3 times with 10 times of to-and pro movement each.

The number of patients required:

We used confidence intervals (CIs) with a prespecified non-inferiority margin of 10% for the non-inferiority analysis. We concluded non-inferiority of PC25 to PC22 if the lower limit of the 95% CI for the difference (PC25-PC22) was not lower than -10%. It was assumed that the diagnostic accuracy of one pass was 75% and that of three cumulative passes was estimated to be 98.4% in PC22. Based on these assumptions, the calculated sample size was 216 samples with power of 80% and significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to participate in research
* 18 years of age and older patients
* Patients who have pancreatic or peripancreatic mass in imaging studies

Exclusion Criteria:

* Contraindication to endoscopy
* Patients younger than 18 years old
* Bleeding tendency
* Cardiopulmonary dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | October. 2014
  Diagnostic accuracy include histologic diAgnosis and cytologic diagnosis

SECONDARY OUTCOMES:
Technical success | October. 2014
  Technical success means the gain of tissue or cells through EUS-guided FNA.

OTHER OUTCOMES:
Complications | November. 2014
  Investigate the occurrence of complications such bleeding and perforation. Not only complications, but the size and location of lesion, puncture routes will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Kwanghyuck Lee, MD, Principal Investigator — Assistant Professor of Medicine, Division of Gastroenterology, Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Seoul City, South Korea